CLINICAL TRIAL: NCT06319677
Title: PK/PD Study of Antibiotics in Critically Ill Patients Receiving ECMO
Brief Title: PK/PD Study of Anti-Infective Drugs in Critically Ill Patients Receiving Extracorporeal Membrane Oxygenation Treatment
Acronym: ECMO
Status: Not yet recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: Ivljingjing
Record Dates: First submitted 2023-09-17; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness; Extracorporeal Membrane Oxygenation Complication
Keywords: Critical Illness; ECMO; Population Pharmacokinetics
MeSH Terms: conditions — Critical Illness | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected before and after dosing according to sampling protocol.Each sample will be about 1-2 mL, for a total of about 12 mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO treatment group: Critically ill adult patients treated with ECMO using one or more antimicrobial agents
  Interventions: Device: ECMO treatment
- Non-ECMO treatment group: Critically ill adult patients using one or more antimicrobial agents not receving ECMO

INTERVENTIONS:
Device: ECMO treatment — Critically ill patients were treated with ECMO while receiving antimicrobial therapy
  Groups: ECMO treatment group

SUMMARY:
Extracorporeal membrane pulmonary oxygenation (ECMO) may provide partial or complete support for organ replacement in patients with severe cardiopulmonary failure, buying time for further management of the primary disease. However, ECMO may significantly alter the pharmacokinetic and pharmacodynamic profiles of critically ill patients, affecting the safety and efficacy of drug therapy. This prospective observational study aims to investigate the impact of ECMO treatment on the pharmacokinetics and pharmacodynamics of antimicrobial drugs in critically ill adult patients. Investigators intend to establish a Population Pharmacokinetic (POP PK) and Pharmacokinetic/Pharmacodynamic (PK/PD) model by prospectively collecting blood samples from patients and relevant treatment data. The primary objective is to quantitatively characterize the pharmacokinetic profiles of critically ill patients undergoing ECMO support and provide model-based recommendations for drug regimens tailored to critically ill patients.

DETAILED DESCRIPTION:
Extracorporeal Membrane Pulmonary Oxygenation (ECMO) is a temporary life-support system used to provide partial or complete organ support for adult patients with severe cardiopulmonary failure. ECMO stabilizes the vital signs of critically ill patients, allowing time for further management of the underlying disease. Effective pharmacologic treatment of the primary condition is crucial for successful patient outcomes.

Critically ill patients often exhibit significant variability in pharmacokinetics (PK) compared to the general population. Moreover, the use of extracorporeal therapeutic techniques like ECMO introduces further variability and unpredictability in drug behavior. This can result from factors such as drug depletion within ECMO circuits, altered drug distribution volumes, and reduced drug excretion.

Sepsis and septic shock due to infections like pneumonia are life-threatening conditions frequently requiring admission to intensive care units. Timely and effective antimicrobial therapy is vital to reduce morbidity and mortality. To investigate the impact of ECMO therapy on the PK and PD of antimicrobial drugs, this prospective observational study will collect blood samples from critically ill adult patients, both those receiving ECMO treatment and those not receiving it. The study will focus on various antimicrobial agents, including imipenem, vancomycin, piperacillin/tazobactam, ceftazidime/avibactam, cefoperazone/sulbactam, cefepime, ceftriaxone, ticlopidine, linezolid, tigecycline, amikacin, gentamicin, polymyxin, voriconazole, fluconazole, caspofungin, micafungin, levofloxacin, and moxifloxacin. Data collected will be used to develop a Population Pharmacokinetic and Pharmacodynamic model based on patient demographics, laboratory results, dosing information, and blood concentration data.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained from the patient or family member
2. Patients who are undergoing ECMO or not
3. Anti-infection treatment indications

Exclusion Criteria:

1. Patients under 18 years of age or pregnant
2. Information on antimicrobial therapy and ECMO support is incomplete
3. Presence of other circumstances that make participation in this study inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients using one or more antimicrobial agents receiving or not receiving ECMO
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Blood drug concentration | Samples were taken in the first 72 hours after administration according to the sampling schedule
  Plasma drug concentration
Pharmacokinetic parameter | 24 hours after administration
  Area under the plasma concentration-time curve（AUC）
Pharmacokinetic parameter | 12 hours after administration
  Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Mortality at 14 and 28 days | Day 30 of the patient's admission
  Mortality was measured by dividing the number of subjects who died during the observation period by the total number of subjects and multiplying by 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Liu, Study Chair — Xiangya Third Hospital, Central South University
Locations (1):
- Xiangya Third Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No